CLINICAL TRIAL: NCT04792879
Title: Assessment of Peripheral Veins Doppler Ultrasound for Diagnosis of Acute Right Heart Failure in Suspicion or Follow-up of Pulmonary Hypertension
Acronym: CODOVEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A00100-41
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Acute Right Heart Failure; Pulmonary Hypertension; Peripheral Veins Doppler Ultrasound
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peripheral veins Doppler ultrasound (Experimental)
  Interventions: Diagnostic Test: Peripheral veins Doppler ultrasound

INTERVENTIONS:
Diagnostic Test: Peripheral veins Doppler ultrasound — Patients undergoing a right heart catheterization for PH diagnosis or annual follow-up in the cardiological unit of the university hospital of Poitiers will be included. A venous Doppler ultrasound will be performed by a vascular physician, with experience in vascular ultrasound imaging, within 4 hours before the right heart catheterization. Morphological parameters of vena cava, and velocimetric parameters of femoral, jugular and supra-hepatic veins will be assessed in order to study their correlation with right auricular pressure value.

SUMMARY:
Occurrence of acute right heart failure (ARHF) remains common during pulmonary hypertension (PH). Right atrial pressure (RAP) invasive measurement is the gold standard to diagnose ARHF in order to improve diuretic treatment management. Existence of indirect signs of ARHF on venous Doppler ultrasound waveform has long been described, but correlation with RAP has not been properly established yet. It is the aim of our study in order to obtain an additional tool to manage ARHF.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 years old)
* Patient referred to the cardiology department for a right heart catheterization with measurement of RAP, regardless of the indication.
* Free subject, without guardianship or curatorship or subordination
* People affiliated to or beneficiary of a social security schemes
* Informed consent signed by the patient after clear and fair information about the study.

Exclusion Criteria:

* Minor patient (age < 18 years)
* Refusal to participate in the study
* Patient with hemodynamic instability, unable to tolerate a delay in treatment caused by the ultrasound examination.
* Patient requiring diuretic treatment within the next 4 hours
* Patient with a life expectancy of less than 24 hours.
* History of proximal deep venous thrombosis involving the inferior vena cava and/or common iliac veins and/or femoral veins.
* History of extrinsic venous compression on the inferior vena cava and/or common iliac veins and/or femoral veins.
* Persons who do not benefit from a Social Security scheme or who do not benefit from it through a third party.
* Persons benefiting from reinforced protection, namely minors, pregnant and nursing women, persons deprived of liberty by a judicial or administrative decision, persons staying in health or social institutions, adults under legal protection and finally patients in emergency situations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive and negative likelihood ratios of venous stasis index | Inclusion day within 4 hours before the right heart catheterization
  Sensitivity, specificity, positive and negative likelihood ratios of venous stasis index*, measured by Pulsed Doppler on common femoral veins, as a diagnostic criterion for ARHF (defined by RAP ≥10 mm Hg).
  * Defined as duration of non-anterograde venous flow during 3 seconds/ 3 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France